CLINICAL TRIAL: NCT07153783
Title: AI-human Collaborative Diagnosis of Liver Tumors Using CE-CT
Brief Title: Interventional AI-Human Collaboration for Liver Tumor Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Deputy director of department of radiology, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SH-CMU-FLL-Intervention
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma (HCC); Intrahepatic Cholangiocarcinoma (Icc); Hepatic Metastasis; Hepatic Hemangioma; Cyst; Focal Nodular Hyperplasia
Keywords: Dynamic Contrast-Enhanced CT; Focal Liver Lesions
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Cysts; Focal Nodular Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-human collaboration in CE-CT diagnosis for liver lesions (Experimental): In the prospective analysis phase, patients undergo routine Multiphasic Contrast-Enhanced Computed Tomography (CE-CT) imaging. The scans are evaluated through two parallel pathways: standard radiologist interpretation (without AI input) and independent AI analysis. When diagnostic discrepancies occur, a senior radiologist or multidisciplinary expert panel reviews the case and provides the definitive diagnosis.
  Interventions: Diagnostic Test: AI-human collaboration for CE-CTs diagnosis

INTERVENTIONS:
Diagnostic Test: AI-human collaboration for CE-CTs diagnosis — The system automatically processes all eligible same-day scans and generates results for review the following day. To maintain efficient AI-human collaboration while preserving the standard clinical workflow, the conventional radiological interpretation process remains unchanged (first-line radiologists provide initial reports followed by senior radiologists' review). A dedicated senior radiologist then evaluates any discordances between AI findings and primary radiological report. For complex cases, the review process escalates to a consensus review panel (i.e., pre-designated senior radiologists, Multidisciplinary Team (MDT)). The MDT can recommend clinical interventions including follow-up (e.g., additional imaging examinations, active surveillance), surgical procedures, or adjustments to adjuvant therapy (initiation or modification of treatment regimens). All discordant cases and their outcomes are systematically documented for longitudinal tracking and follow-up analysis.

SUMMARY:
Recent advances in artificial intelligence (AI), particularly deep learning technology, have transformed medical imaging analysis. AI systems have demonstrated diagnostic performance comparable to or exceeding that of expert radiologists in specific tasks. Liver-focused AI diagnostic systems have achieved promising results in multi-center validations; however, these retrospective studies have not yet addressed two critical gaps. First, large-scale prospective trials are required to establish real-world clinical effectiveness. Second, it remains unclear whether AI can be organically embedded into clinical diagnostic workflows to reshape diagnostic and therapeutic pathways, particularly by enhancing the detection and follow-up of hepatic malignancies and ultimately improving patient outcomes.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of AI-human collaboration in liver tumor diagnosis by embedding real-time AI analysis into conventional multiphasic contrast-enhanced CT (CE-CT) workflows. Specifically, this prospective validation trial will assess diagnostic performance in detecting and characterizing hepatic lesions, particularly malignancies, evaluate the feasibility and efficiency of workflow integration, and determine the potential clinical impact on treatment decision-making and patient management.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18 years and above
2. Underwent dynamic contrast-enhanced abdominal CT examination with liver coverage
3. Imaging must include at least three required phases: non-contrast, arterial phase, and venous phase; an delayed phase is optional
4. Complete imaging data that meet AI system analysis requirements.

Exclusion Criteria:

1. History of recent upper-abdominal surgery (within 30 days) or major hepatobiliary-pancreatic surgery affecting liver evaluation (e.g., liver transplantation or Whipple procedure); patients with prior simple cholecystectomy or single-lesion interventional procedures are not excluded
2. History of recent hepatic trauma (within 30 days)
3. Poor image quality or severe noise artifacts (e.g., metal or motion artifacts)
4. Missing required imaging phases (required at least non-contrast, arterial, and venous phases) or inadequate scan range (e.g., lower-abdomen CT such as pelvic or rectal scans not covering the liver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10333 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the AI System for malignancy diagnosis | Up to 90 days
  Measures the patient-level diagnostic accuracy of the AI system for differentiating malignant vs. non-malignant lesions. The primary metric is the Area under the Receiver Operating Characteristic Curve (AUC). The primary analysis will test the one-sided superiority hypothesis H1: AUC > 0.90 against H0: AUC <= 0.90. The trial will be considered successful if the lower bound of the 95% Confidence Interval (CI) for the AUC is greater than 0.90.

SECONDARY OUTCOMES:
Secondary diagnostic performance | Up to 90 days
  Measures the patient-level diagnostic performance of the AI system for malignant versus non-malignant classification. Metrics include sensitivity, specificity, Positive Predictive Value (PPV), and Negative Predictive Value (NPV). These will be calculated from the continuous probability score using a fixed operating point prior to prospective analysis.
Lesion screening performance | Up to 90 days
  Measures the patient-level screening ability of the AI system to distinguish patients with any lesion from those with no lesions. This is a binary classification task (AUC) comparing lesion patient (malignant or benign) versus no lesion (normal liver or diffuse disease only).
Detection discordance | Up to 90 days
  Measures the number of FLLs identified by the AI-human collaborative workflow that were overlooked by the initial radiologist report. An overlooked lesion is defined as an event meeting all three criteria: (1) detected by the AI system; (2) not described in the initial radiological report; (3) confirmed as a true lesion by senior radiologist/MDT re-review.
Amended radiological report | Up to 90 days
  Measures the number of formal addenda issued to finalized radiology reports. An amended report is defined as a formal addendum that explicitly corrects a diagnosis or adds a previously missed finding based on the AI-human collaborative review.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, MD PhD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share IPD related to abdominal dynamic-contrast enhanced CT scans and clinical outcomes for hepatic tumor diagnosis.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Ding W, Meng Y, Ma J, Pang C, Wu J, Tian J, Yu J, Liang P, Wang K. Contrast-enhanced ultrasound-based AI model for multi-classification of focal liver lesions. J Hepatol. 2025 Aug;83(2):426-439. doi: 10.1016/j.jhep.2025.01.011. Epub 2025 Jan 21. PMID 39848548
- [Background] Ying H, Liu X, Zhang M, Ren Y, Zhen S, Wang X, Liu B, Hu P, Duan L, Cai M, Jiang M, Cheng X, Gong X, Jiang H, Jiang J, Zheng J, Zhu K, Zhou W, Lu B, Zhou H, Shen Y, Du J, Ying M, Hong Q, Mo J, Li J, Ye G, Zhang S, Hu H, Sun J, Liu H, Li Y, Xu X, Bai H, Wang S, Cheng X, Xu X, Jiao L, Yu R, Lau WY, Yu Y, Cai X. A multicenter clinical AI system study for detection and diagnosis of focal liver lesions. Nat Commun. 2024 Feb 7;15(1):1131. doi: 10.1038/s41467-024-45325-9. PMID 38326351
- [Background] Cao K, Xia Y, Yao J, Han X, Lambert L, Zhang T, Tang W, Jin G, Jiang H, Fang X, Nogues I, Li X, Guo W, Wang Y, Fang W, Qiu M, Hou Y, Kovarnik T, Vocka M, Lu Y, Chen Y, Chen X, Liu Z, Zhou J, Xie C, Zhang R, Lu H, Hager GD, Yuille AL, Lu L, Shao C, Shi Y, Zhang Q, Liang T, Zhang L, Lu J. Large-scale pancreatic cancer detection via non-contrast CT and deep learning. Nat Med. 2023 Dec;29(12):3033-3043. doi: 10.1038/s41591-023-02640-w. Epub 2023 Nov 20. PMID 37985692